CLINICAL TRIAL: NCT06455813
Title: Oral Laxatives After Hip Fracture Surgery: A Randomised Controlled Trial
Brief Title: What Laxative Should be Used After Hip Fracture Surgery?
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Independent Research Fund Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Laxatives26092019
Record Dates: First submitted 2024-05-03; First posted 2024-06-12 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Bisacodyl; polyethylene glycol 3350; Electrolytes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Macrogol 3350 and electrolytes. (Active Comparator): Powder for oral solution in sachet Macrogol 3350 and electrolytes (ATC code A06AD65) which is administered orally as the content of 2 sachets daily (in the evening) during admission
  Interventions: Drug: Macrogol 3350 and electrolytes
- Bisacodyl (Active Comparator): Enteric coated tablet Bisacodyl (ATC code A06AB02) 5 mg, 2 tablets daily which is administered orally daily (in the evening) during admission
  Interventions: Drug: Bisacodyl
- A combination of macrogol 3350 and electrolytes and bisacodyl (Active Comparator): Powder for oral solution in sachet macrogol 3350 and electrolytes (ATC code A06AD65) which is administered orally daily (in the evening) as the content of 1 sachet given in combination with enteric coated tablet Bisacodyl (ATC code A06AB02) 5 mg, 1 tablet orally daily (in the evening) during admission
  Interventions: Drug: A combination of macrogol 3350 and electrolytes and bisacodyl

INTERVENTIONS:
Drug: Bisacodyl — The patients' stool frequency, degree of constipation and side effects of the medication as well as pain, nausea and flatulence are scored once a day using the Bristol Stool Scale, Verbal Rank Scale and Patient Assessment of Constipation symptoms Questionnaire. If the first defecation has not occurred 72 hours after the end of the operation, the patients in all three groups are transferred to treatment with peristaltic-promoting agents
  Other Names: Dulcolax
  Arms: Bisacodyl
Drug: Macrogol 3350 and electrolytes — The patients' stool frequency, degree of constipation and side effects of the medication as well as pain, nausea and flatulence are scored once a day using the Bristol Stool Scale, Verbal Rank Scale and Patient Assessment of Constipation symptoms Questionnaire. If the first defecation has not occurred 72 hours after the end of the operation, the patients in all three groups are transferred to treatment with peristaltic-promoting agents
  Other Names: Gangiden
  Arms: Macrogol 3350 and electrolytes.
Drug: A combination of macrogol 3350 and electrolytes and bisacodyl — The patients' stool frequency, degree of constipation and side effects of the medication as well as pain, nausea and flatulence are scored once a day using the Bristol Stool Scale, Verbal Rank Scale and Patient Assessment of Constipation symptoms Questionnaire. If the first defecation has not occurred 72 hours after the end of the operation, the patients in all three groups are transferred to treatment with peristaltic-promoting agents
  Other Names: A combination of Gangiden og Dulcolax
  Arms: A combination of macrogol 3350 and electrolytes and bisacodyl

SUMMARY:
To conduct a randomized clinical trial to determine how best to prevent constipation after hip fracture surgery using laxatives.

DETAILED DESCRIPTION:
Background:

Acute constipation is very common in connection with major operations. Constipation is a complication that can prolong hospital stays, increase nursing time and healthcare costs. Up to 70% experience constipation after surgery for a hip fracture. Prevention of constipation is considered an important part of treatment after hip surgery, but although the use of anti-constipation drugs is widespread, there are no studies of sufficient quality to show how and with what means constipation is best treated. For the same reason, in Denmark there is great variation in the approach to preventive treatment - and thus also the treatment result.

Aim:

The aim is to investigate how to prevent constipation best after hip surgery using laxatives.

Method, design, intervention og investigation procedures:

The project is a randomized controlled trial in ratio 1:1:1, where the patients assigned to two different orthopedic surgery departments are assigned to either have one of two drugs (bisacodyl, macrogol) or both types of anti-constipation drugs. It is calculated that 375 patients will be included in the trial, i.e. 125 patients in each group. It is expected that patients will be evenly included distributed between two hospitals.

The patients will respectively be given macrogol 3350 and electrolytes (ATC code A06AD65) which is administered as the content of 2 sachets, Bisacodyl (ATC code A06AB02) 5 mg, 2 tablets or a combination of both in half the dose.

All laxatives are administered orally in the evening on the day of surgery (the next standard administration time at 10 pm) and it is known to both patients and staff which trial medication each patient is receiving. The patients' stool frequency, degree of constipation and side effects of the medication as well as pain, nausea and flatulence are scored once a day using the Bristol Stool Scale, Verbal Rank Scale and Patient Assessment of Constipation symptoms Questionnaire. If the first defecation has not occurred 72 hours after the end of the operation, the patients in all three groups are transferred to treatment with peristalsis-promoting agents Bisacodyl 5 mg, 2 tablets. The patients stay in the trial and get the trial medication they are assigned to unless an orthopedic surgeon assesses otherwise.

ELIGIBILITY:
Inclusion Criteria:

* Acute hip fracture surgery patients from one of two orthopedic departments from hospitals in the Southern Region of Denmark.
* Age≥ 65 years
* The patients should be able to speak and understand Danish.

Exclusion Criteria:

* Patients:

  * with known chronic constipation (defined from Wexner constipation score)
  * with known use of laxatives at admission
  * who participate in other similar clinical studies
  * who is terminally ill
  * who is restraint
  * who is in isolation
  * with severe heart disease defined as New York Heart Association (NYHA) III og IV
  * with severe chronically inflammatory bowel disease
  * with acute abdominal surgical conditions, eg. ileus, obstruction or perforation
  * with dysphagia where the patient can not swallow tablets/oral liquids
  * with toxic megacolon
  * with gastric emptying disorder
  * with severe electrolyte disorder (P-kalium: < 2.5 mmol/l og P-natrium: <125 mmol/l)
  * Allergies to the ingredients
  * Pregnant women can not be included but the women are expected to be postmenopausal why pregnancy test are not performed

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who will need rescue medication (Bisacodyl) | 72 hours after surgery
  Part of patients in each group who needs rescue medication after 72 hours or rescue medication before 72 hours on behalf of a medical assessment

SECONDARY OUTCOMES:
Time to first bowel movements | hours up to 240 hours
  Time to first bowel movements (in hours after finished surgery)
Length of hospital stay | days up to 10 days
  Length of hospital stay of the index admission from admission to discharge
Number of patients who are readmitted at hospital | 30 days
  The part of patients who are readmitted at hospital 30 days after discharge hospital
Number of patients who have emergency room visits | 30 days
  The proportion of patients who have emergency room visits within 30 days of discharge hospital
Constipation defined from the Bristol Stool Scale | daily up to 10 days
  constipation defined from the Bristol Stool Scale with type 1-7 where type 1 is constipation and type 7 is diarrhea and use/no use of rescue medication (bisacodyl)
Constipation score | daily up to 10 days
  Calculated score based of The Patient Assessment of Constipation symptoms Questionnaire from 0-48 where 48 is most severe constipation and use/no use of rescue medication (bisacodyl)

CONTACTS AND LOCATIONS:
Overall Officials: Carina Lundby, Study Director — Odense University Hospital
Locations (2):
- Denmark (2):
  - Hospital Lillebælt, Kolding Hospital, Kolding
  - Odense University Hospital, Svendborg Hospital, Svendborg

IPD SHARING:
Plan to Share IPD: No